CLINICAL TRIAL: NCT01399879
Title: Measuring Skin Electrical Potential With the Kelvin Probe: Minimizing Noise
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Andrew C. Ahn, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 5R21AT005249 (NIH)
Record Dates: First submitted 2011-03-25; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Healthy State
Keywords: Surface potential; Electrical; Motion stabilization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers
  Interventions: Other: Faraday cage, movement stabilization

INTERVENTIONS:
Other: Faraday cage, movement stabilization — The Faraday cage is a copper-mesh cage that surrounds the device and test site. It helps eliminate surrounding electrical noise. Movement stabilization will be achieved by placing a velcro strap over the arm to minimize random movements.

SUMMARY:
The Scanning Kelvin Probe measures surface electrical potential without actually touching the skin. This is a pilot study to evaluate methods of minimizing noise during Scanning Kelvin Probe measurements. This project will focus specifically on noise arising from physical movement and environmental electrical field.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years

Exclusion Criteria:

* chronic medical condition requiring daily medications (hypertension, diabetes, hypothyroidism, etc)
* movement disorders/tremors
* extensive scars on the hand
* latex-allergies
* cardiac implantation, metallic joint/bone replacements (defibrillator or pacemaker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Variability in surface electrical potential measurements | Within 24 hours of testing
  This study focuses on the ability of the Kelvin Probe to measure skin electrical potential. Because it does so without touching the skin, it is prone to noise - specifically physical movement and surrounding electrical noise. The variability in surface electrical potential is a way to determine how stable the measurements are. It can be determined immediately after testing - and will be used in data analyses (comparing across study volunteers) approximately 24 weeks after testing is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Ahn, MD MPH, Principal Investigator — Massachusetts General Hospital